CLINICAL TRIAL: NCT02630108
Title: Clinical Study of Transarterial Chemoembolization (TACE) Combined With Synchronous Radiofrequency /Microwave Ablation to Treat Large and Huge Hepatocellular Carcinoma
Brief Title: TACE Combined With Synchronous Radiofrequency /Microwave Ablation to Treat Large and Huge Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Xijing Hospital (Other); Changhai Hospital (Other); Eastern Hepatobiliary Surgery Hospital (Other); Shanghai Cancer Hospital, China (Other); Shengjing Hospital (Other); The Third Affiliated Hospital of Harbin Medical University (Other); Jilin Provincial Tumor Hospital (Other); Zhejiang Cancer Hospital (Other); Jiangsu Cancer Institute & Hospital (Other); Guangdong Provincial People's Hospital (Other); Sichuan Cancer Hospital and Research Institute (Other); Henan Cancer Hospital (Other Government); Anhui Provincial Hospital (Other Government); The First Affiliated Hospital of Anhui Medical University (Other); Qilu Hospital of Shandong University (Other); Shandong Tumor Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Chinese PLA General Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); LanZhou University (Other); Sun Yat-sen University (Other); Hunan Provincial People's Hospital (Other); Affiliated Zhongshan Hospital of Dalian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2015-146R
Record Dates: First submitted 2015-12-03; First posted 2015-12-15 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Carcinoma, Hepatocellular
Keywords: HCC; TACE; Thermal Ablation; Safety/Efficacy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Transurethral Resection of Prostate; Radiofrequency Ablation; Epirubicin; Ethiodized Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thermal Ablation & TACE (Experimental): Transarterial chemoembolization (TACE) is performed immediately following thermal ablation.
  EADM, ultra-fluid lipiodol and gelatin sponge articles are used in TACE.
  Interventions: Procedure: Thermal Ablation; Drug: EADM; Drug: Ultra-fluid lipiodol; Other: Gelatin sponge articles
- TACE alone (Active Comparator): Only TACE is performed. EADM, ultra-fluid lipiodol and gelatin sponge articles are used in TACE.
  Interventions: Drug: EADM; Drug: Ultra-fluid lipiodol; Other: Gelatin sponge articles

INTERVENTIONS:
Procedure: Thermal Ablation — Thermal ablation in this trial includes radiofrequency ablation and microwave ablation, one of them can be chosen to be performed.
  Other Names: Radiofrequency ablation; Microwave ablation
  Arms: Thermal Ablation & TACE
Drug: EADM — EADM is a chemotherapy drug used in transarterial chemoembolization (TACE).Dosage: EADM 30-60 mg per patient,depending on the situation of the patient.
  Other Names: Epirubicin
Drug: Ultra-fluid lipiodol — Ultra-fluid lipiodol is a kind of embolization material used in TACE. Standard: 38% ultra-fluid lipiodol .
  Other Names: lipiodol
Other: Gelatin sponge articles — Gelatin sponge articles embolization material used in TACE. Standard: 350-560 um in diameter.

SUMMARY:
It is a prospective and multi-center clinical research in China to compare the efficacy, safety and related impact factors between TACE alone and TACE combined with synchronous multi-point MWA/RFA for large and huge liver cancer.

DETAILED DESCRIPTION:
It is an open random prospective phase III clinical trial conducted by Principal Investigator Professor Jian-Hua Wang. Investigators in twenty-five hospitals in China participate in. Patients with unresectable large HCC (>5cm in diameter) and huge HCC (>=10cm in diameter) are enrolled. The investigators propose to recruitment 280 patients who are randomly assigned into the combined group (treated with TACE and synchronous ablation) and the control group (treated with TACE alone) according to the proportion of 1:1, which means 140 patients in each group. The criteria of inclusion and exclusion, and the methods of lab tests, imaging modality and treatment procedures are the same.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary liver cancer aged from 18-80 years, and life expectancy longer than three months;
2. Patients with large HCC (>5cm in diameter) and huge HCC (≥10cm in diameter), including HCC and mixed type of liver cancer (HCC-ICC);
3. Patients with no thrombus in main portal vein (PV)
4. Patients' liver function classified as Child-Pugh A or B, ECOG PS ≤ 2;
5. Patients without bleeding tendency or coagulation disorder, or with reversible coagulopathy after therapy;
6. White blood cell count ≥ 3.0×10^9/L;
7. Hemoglobin ≥ 8.5g/dl;
8. Platelet ≥ 50×10^9/L;
9. INR ≤ 2.3 or PT not exceeding the upper limit of reference 3 seconds;
10. Blood creatinine less than 1.5 times of upper limit of reference;
11. Patients and/or their relatives willing to join in the clinical trial and signing the informed consent.

Exclusion Criteria:

1. Patients with diffuse type of liver cancer;
2. Cholangiocellular carcinoma
3. Patients with main PV thrombus;
4. Patients with hepatic vein thrombus;
5. Patients with lymph node or distant metastasis outside of liver;
6. Patients' liver function classified as Child-Pugh C and no improvement after treatment of liver protection;
7. Patients with irreversible coagulation disorder and abnormality in blood routine test, or having obvious bleeding tendency;
8. Patients with intractable massive ascites;
9. Patients' ECOG PS >2;
10. Patients complicated with active infection, especially cholangitis;
11. Patients with severe disorders of heart, lungs, kidneys, or brain;
12. Patients and/or their relatives refuse to anticipate this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From the date of randomization until the date of death from any cause, assessed up to 26 months

SECONDARY OUTCOMES:
Time-to-Disease Progression | From the date of first procedure of TACE or TACE combined with synchronous ablation until the time when the disease progresses from an intermediate to an advanced stage as defined by specific events, assessed up to 26 months
  TTDP follow-up is done at three months interval after lesions defined as stable with treatment of TACE or ablation combined with synchronous TACE six months after enrollment until lesions are defined as disease progression.
Objective response rate (ORR) | Six months after the date of first procedure of TACE or TACE combined with synchronous ablation.
  The ratio of CR plus PR. The efficacy is defined as complete regression (CR), partial regression (PR), stable disease (SD) and progressive disease (PD) according to modified Response Evaluation Criteria in Solid Tumors (mRESIST)
Progression free survival(PFS) | From the date of first procedure of TACE or TACE combined with synchronous ablationto until the time when lesions are defined as disease progression or death by any cause,assessed up to 26 months.
Numbers of TACE and TACE combined with ablation cycles | From the date of randomization until the date of death, assessed up to 26 months.
  The times of the subjects undergoing TACE or TACE combined with ablation
Number of participants with adverse events and severe adverse events in TACE alone and TACE combined with ablation groups | From the date of randomization until the date of follow-up visit (30 days after the procedure of TACE or TACE combined with thermal ablation)
  Serious or mild adverse events after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Wang, MD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Department of Interventional Radiology, Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2015. CA Cancer J Clin. 2015 Jan-Feb;65(1):5-29. doi: 10.3322/caac.21254. Epub 2015 Jan 5. PMID 25559415
- [Result] Forner A, Llovet JM, Bruix J. Hepatocellular carcinoma. Lancet. 2012 Mar 31;379(9822):1245-55. doi: 10.1016/S0140-6736(11)61347-0. Epub 2012 Feb 20. PMID 22353262
- [Result] Zhang L, Yin X, Gan YH, Zhang BH, Zhang JB, Chen Y, Xie XY, Ge NL, Wang YH, Ye SL, Ren ZG. Radiofrequency ablation following first-line transarterial chemoembolization for patients with unresectable hepatocellular carcinoma beyond the Milan criteria. BMC Gastroenterol. 2014 Jan 10;14:11. doi: 10.1186/1471-230X-14-11. PMID 24410841
- [Result] Mabed M, Esmaeel M, El-Khodary T, Awad M, Amer T. A randomized controlled trial of transcatheter arterial chemoembolization with lipiodol, doxorubicin and cisplatin versus intravenous doxorubicin for patients with unresectable hepatocellular carcinoma. Eur J Cancer Care (Engl). 2009 Sep;18(5):492-9. doi: 10.1111/j.1365-2354.2008.00984.x. PMID 19453695
- [Result] Llovet JM, Real MI, Montana X, Planas R, Coll S, Aponte J, Ayuso C, Sala M, Muchart J, Sola R, Rodes J, Bruix J; Barcelona Liver Cancer Group. Arterial embolisation or chemoembolisation versus symptomatic treatment in patients with unresectable hepatocellular carcinoma: a randomised controlled trial. Lancet. 2002 May 18;359(9319):1734-9. doi: 10.1016/S0140-6736(02)08649-X. PMID 12049862
- [Result] Koo JE, Kim JH, Lim YS, Park SJ, Won HJ, Sung KB, Suh DJ. Combination of transarterial chemoembolization and three-dimensional conformal radiotherapy for hepatocellular carcinoma with inferior vena cava tumor thrombus. Int J Radiat Oncol Biol Phys. 2010 Sep 1;78(1):180-7. doi: 10.1016/j.ijrobp.2009.07.1730. Epub 2009 Nov 18. PMID 19926229
- [Result] Shiomi H, Naka S, Sato K, Demura K, Murakami K, Shimizu T, Morikawa S, Kurumi Y, Tani T. Thoracoscopy-assisted magnetic resonance guided microwave coagulation therapy for hepatic tumors. Am J Surg. 2008 Jun;195(6):854-60. doi: 10.1016/j.amjsurg.2007.08.056. Epub 2008 Mar 26. PMID 18355796
- [Result] Liu C, Liang P, Liu F, Wang Y, Li X, Han Z, Liu C. MWA combined with TACE as a combined therapy for unresectable large-sized hepotocellular carcinoma. Int J Hyperthermia. 2011;27(7):654-62. doi: 10.3109/02656736.2011.605099. Epub 2011 Oct 3. PMID 21966941
- [Result] Gillams A. Tumour ablation: current role in the liver, kidney, lung and bone. Cancer Imaging. 2008 Oct 4;8 Spec No A(Spec Iss A):S1-5. doi: 10.1102/1470-7330.2008.9001. PMID 18852074
- [Result] Livraghi T, Goldberg SN, Lazzaroni S, Meloni F, Solbiati L, Gazelle GS. Small hepatocellular carcinoma: treatment with radio-frequency ablation versus ethanol injection. Radiology. 1999 Mar;210(3):655-61. doi: 10.1148/radiology.210.3.r99fe40655. PMID 10207464
- [Result] Goldberg SN, Charboneau JW, Dodd GD 3rd, Dupuy DE, Gervais DA, Gillams AR, Kane RA, Lee FT Jr, Livraghi T, McGahan JP, Rhim H, Silverman SG, Solbiati L, Vogl TJ, Wood BJ; International Working Group on Image-Guided Tumor Ablation. Image-guided tumor ablation: proposal for standardization of terms and reporting criteria. Radiology. 2003 Aug;228(2):335-45. doi: 10.1148/radiol.2282021787. PMID 12893895
- [Result] Gillams AR. Image guided tumour ablation. Cancer Imaging. 2005 Sep 21;5(1):103-9. doi: 10.1102/1470-7330.2005.0015. PMID 16305946
- [Result] Ito A, Shinkai M, Honda H, Yoshikawa K, Saga S, Wakabayashi T, Yoshida J, Kobayashi T. Heat shock protein 70 expression induces antitumor immunity during intracellular hyperthermia using magnetite nanoparticles. Cancer Immunol Immunother. 2003 Feb;52(2):80-8. doi: 10.1007/s00262-002-0335-x. Epub 2003 Jan 29. PMID 12594571
- [Result] Dong BW, Zhang J, Liang P, Yu XL, Su L, Yu DJ, Ji XL, Yu G. Sequential pathological and immunologic analysis of percutaneous microwave coagulation therapy of hepatocellular carcinoma. Int J Hyperthermia. 2003 Mar-Apr;19(2):119-33. doi: 10.1080/0265673021000017154. PMID 12623635
- [Result] Xu LF, Sun HL, Chen YT, Ni JY, Chen D, Luo JH, Zhou JX, Hu RM, Tan QY. Large primary hepatocellular carcinoma: transarterial chemoembolization monotherapy versus combined transarterial chemoembolization-percutaneous microwave coagulation therapy. J Gastroenterol Hepatol. 2013 Mar;28(3):456-63. doi: 10.1111/jgh.12088. PMID 23216261
- [Result] Cross FA, Evans DW, Barber RT. Decadal Declines of Mercury in Adult Bluefish (1972-2011) from the Mid-Atlantic Coast of the U.S.A. Environ Sci Technol. 2015 Aug 4;49(15):9064-72. doi: 10.1021/acs.est.5b01953. Epub 2015 Jul 21. PMID 26148053
- [Result] Lencioni R, Llovet JM. Modified RECIST (mRECIST) assessment for hepatocellular carcinoma. Semin Liver Dis. 2010 Feb;30(1):52-60. doi: 10.1055/s-0030-1247132. Epub 2010 Feb 19. PMID 20175033
- [Result] Takayasu K, Arii S, Kudo M, Ichida T, Matsui O, Izumi N, Matsuyama Y, Sakamoto M, Nakashima O, Ku Y, Kokudo N, Makuuchi M. Superselective transarterial chemoembolization for hepatocellular carcinoma. Validation of treatment algorithm proposed by Japanese guidelines. J Hepatol. 2012 Apr;56(4):886-92. doi: 10.1016/j.jhep.2011.10.021. Epub 2011 Dec 13. PMID 22173160
- [Result] Terzi E, Piscaglia F, Forlani L, Mosconi C, Renzulli M, Bolondi L, Golfieri R; BLOG-Bologna Liver Oncology Group, S.Orsola-Malpighi Hospital, University of Bologna, Bologna, Italy. TACE performed in patients with a single nodule of hepatocellular carcinoma. BMC Cancer. 2014 Aug 19;14:601. doi: 10.1186/1471-2407-14-601. PMID 25139639
- [Result] Lencioni R, Crocetti L. Local-regional treatment of hepatocellular carcinoma. Radiology. 2012 Jan;262(1):43-58. doi: 10.1148/radiol.11110144. PMID 22190656
- [Result] Goldberg SN, Grassi CJ, Cardella JF, Charboneau JW, Dodd GD 3rd, Dupuy DE, Gervais DA, Gillams AR, Kane RA, Lee FT Jr, Livraghi T, McGahan J, Phillips DA, Rhim H, Silverman SG, Solbiati L, Vogl TJ, Wood BJ, Vedantham S, Sacks D; Society of Interventional Radiology Technology Assessment Committee and the International Working Group on Image-guided Tumor Ablation. Image-guided tumor ablation: standardization of terminology and reporting criteria. J Vasc Interv Radiol. 2009 Jul;20(7 Suppl):S377-90. doi: 10.1016/j.jvir.2009.04.011. PMID 19560026
- [Result] Qian GJ, Wang N, Shen Q, Sheng YH, Zhao JQ, Kuang M, Liu GJ, Wu MC. Efficacy of microwave versus radiofrequency ablation for treatment of small hepatocellular carcinoma: experimental and clinical studies. Eur Radiol. 2012 Sep;22(9):1983-90. doi: 10.1007/s00330-012-2442-1. Epub 2012 Apr 28. PMID 22544225
- [Result] Abdelaziz A, Elbaz T, Shousha HI, Mahmoud S, Ibrahim M, Abdelmaksoud A, Nabeel M. Efficacy and survival analysis of percutaneous radiofrequency versus microwave ablation for hepatocellular carcinoma: an Egyptian multidisciplinary clinic experience. Surg Endosc. 2014 Dec;28(12):3429-34. doi: 10.1007/s00464-014-3617-4. Epub 2014 Jun 17. PMID 24935203
- [Result] Poggi G, Montagna B, DI Cesare P, Riva G, Bernardo G, Mazzucco M, Riccardi A. Microwave ablation of hepatocellular carcinoma using a new percutaneous device: preliminary results. Anticancer Res. 2013 Mar;33(3):1221-7. PMID 23482806
- [Result] Liu Y, Zheng Y, Li S, Li B, Zhang Y, Yuan Y. Percutaneous microwave ablation of larger hepatocellular carcinoma. Clin Radiol. 2013 Jan;68(1):21-6. doi: 10.1016/j.crad.2012.05.007. Epub 2012 Jul 4. PMID 22766484
- [Result] Ni JY, Sun HL, Chen YT, Luo JH, Chen D, Jiang XY, Xu LF. Prognostic factors for survival after transarterial chemoembolization combined with microwave ablation for hepatocellular carcinoma. World J Gastroenterol. 2014 Dec 14;20(46):17483-90. doi: 10.3748/wjg.v20.i46.17483. PMID 25516662
- [Result] Yin XY, Xie XY, Lu MD, Xu HX, Xu ZF, Kuang M, Liu GJ, Liang JY, Lau WY. Percutaneous thermal ablation of medium and large hepatocellular carcinoma: long-term outcome and prognostic factors. Cancer. 2009 May 1;115(9):1914-23. doi: 10.1002/cncr.24196. PMID 19241423
- [Result] Forner A, Real MI, Varela M, Bruix J. Transarterial chemoembolization for patients with hepatocellular carcinoma. Hepatol Res. 2007 Sep;37 Suppl 2:S230-7. doi: 10.1111/j.1872-034X.2007.00190.x. PMID 17877488
- [Result] Liang P, Wang Y, Yu X, Dong B. Malignant liver tumors: treatment with percutaneous microwave ablation--complications among cohort of 1136 patients. Radiology. 2009 Jun;251(3):933-40. doi: 10.1148/radiol.2513081740. Epub 2009 Mar 20. PMID 19304921
- [Result] Ding J, Jing X, Liu J, Wang Y, Wang F, Wang Y, Du Z. Complications of thermal ablation of hepatic tumours: comparison of radiofrequency and microwave ablative techniques. Clin Radiol. 2013 Jun;68(6):608-15. doi: 10.1016/j.crad.2012.12.008. Epub 2013 Feb 8. PMID 23399463
- See also: Link Text:BioMed Central — http://www.biomedcentral.com/content/pdf/1471-230X-14-11.pdf
- See also: Link Text:Wiley — http://onlinelibrary.wiley.com/doi/10.1111/j.1365-2354.2008.00984.x/pdf
- See also: Link Text:PubMed Central — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2582496/pdf/ci089001.pdf
- See also: Link Text:PubMed Central — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC1665233/pdf/ci050103.pdf
- See also: Link Text:ProQuest Health and Medical Complete New Platform — http://search.proquest.com/docview/213492101?accountid=10025
- See also: Link Text:Wiley — http://onlinelibrary.wiley.com/doi/10.1111/jgh.12088/epdf
- See also: Link Text:Georg Thieme Verlag Stuttgart, New York — https://www.thieme-connect.com/products/ejournals/html/10.1055/s-0030-1247132
- See also: Link Text:BioMed Central — http://www.biomedcentral.com/content/pdf/1471-2407-14-601.pdf
- See also: Link Text:Link Text: — http://pubs.rsna.org/doi/10.1148/radiol.11110144?url_ver=Z39.88-2003&rfr_id=ori:rid:crossref.org&rfr_dat=cr_pub%3dpubmed
- See also: Link Text:ProQuest Health and Medical Complete New Platform — http://search.proquest.com/docview/1032640168?accountid=10025
- See also: Link Text:Springer — http://link.springer.com/content/pdf/10.1007%2Fs00464-014-3617-4.pdf
- See also: Link Text:HighWire — http://ar.iiarjournals.org/content/33/3/1221.full.pdf+html
- See also: Link Text:Wiley — http://onlinelibrary.wiley.com/doi/10.1002/cncr.24196/pdf